CLINICAL TRIAL: NCT06672835
Title: Beliefs and Attitudes for Successful Implementation in Schools (BASIS) Optimization
Brief Title: BASIS Optimization
Acronym: BASIS R34
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Kansas (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Lyon, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00021393; 5P50MH126219-04 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Health Services; Evidence Based Programs in Schools
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention study model is parallel where participants will be randomly assigned to the experimental group (n=16) and the active comparator group (n=16).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eBASIS (Experimental): eBASIS is an online, optimized, and evidence-based practice agnostic implementation strategy that addresses the behavioral component often missing from standard evidence-based practice training and consultation. It relates to motivation before and volition after the evidence-based practice training and targets behavioral intentions by improving attitudes, subjective norms, and self-efficacy. The implementation strategy is designed to be designed to be delivered within the Preparation/Adoption phase immediately prior to the Action implementation in the EPIS model.
  Interventions: Behavioral: eBASIS
- eAttention Control (Placebo Comparator): eAC is an online control for eBASIS. Providers assigned to eAttention Control (eAC) will receive pre- and post-training experiences designed to mirror those received in eBASIS. These training experiences will be delivered on the same platform and be approximately the same length as the eBASIS but will not contain any eBASIS content or mechanisms of change. The eAC pre-training experience will define, describe, and advocate for evidence-based practice implementation in schools. Content in eAC will be didactic similar to a typical professional development training for providers.
  Interventions: Behavioral: eAttention Control

INTERVENTIONS:
Behavioral: eBASIS — eBASIS is an online, optimized, and evidence-based practice agnostic implementation strategy that addresses the behavioral component often missing from standard evidence-based practice training and consultation. It relates to motivation before and volition after the evidence-based practice training and targets behavioral intentions by improving attitudes, subjective norms, and self-efficacy. The implementation strategy is designed to be designed to be delivered within the Preparation/Adoption phase immediately prior to the Action implementation in the EPIS model.
  Arms: eBASIS
Behavioral: eAttention Control — eAC is an online control for eBASIS. Providers assigned to eAttention Control (eAC) will receive pre- and post-training experiences designed to mirror those received in eBASIS. These training experiences will be delivered on the same platform and be approximately the same length as the eBASIS but will not contain any eBASIS content or mechanisms of change. The eAC pre-training experience will define, describe, and advocate for evidence-based practice implementation in schools. Content in eAC will be didactic similar to a typical professional development training for providers.
  Arms: eAttention Control

SUMMARY:
The objective of the BASIS R34 pilot study is to test the impact of eBASIS in a randomized controlled trial (RCT). Consistent with IMPACT's IQM, the study tests effects of eBASIS on treatment fidelity and youth outcomes, compared to a digitally delivered control (N=32 clinicians; 96 clients). A well-established EBP (Cognitive Behavioral Therapy Plus), will be a focus of the investigation, which eligible participants will already be signed up to receive.

DETAILED DESCRIPTION:
Although evidence-based practices (EBPs) have been extensively developed, they are not widely used in school settings, where up to 80% of youth receive mental health services. This results in reduced impact on youth mental health. The project aims to test the online version of efficient and effective strategy called BASIS to improve the quality of EBP by focusing on individual-level processes, complementing organizational change approaches.

The strategy applies the Theory of Planned Behavior (TPB) to influence key provider behaviors, such as attitudes, subjective norms, and perceived behavioral control, which are central to EBP adoption and fidelity. Preliminary trials on BASIS found significant changes in key theory of planned behavior mechanisms (e.g., attitudes, perceived behavioral control, and social norms) and more engagement in post-training consultation among school school-based clinicians, supporting implementation of evidenced-based social-emotional-behavioral practices. By addressing the intrapersonal mechanisms driving provider decisions, the study aims to improve implementation outcomes in school settings.

The objective of this pilot study is to test the impact of the optimized eBASIS in a randomized controlled trial (RCT). Consistent with IMPACT's IQM, the study tests effects of eBASIS on treatment fidelity and youth outcomes, compared to a digitally delivered control (N=32 clinicians; 96 clients). A well-established EBP (Cognitive Behavioral Therapy Plus), will be a focus of the investigation, which eligible participants will already be signed up to receive.

ELIGIBILITY:
Inclusion Criteria:

* Mental health provider who spends 2 hours or more providing supports in school setting
* Registered to receive CBT+ training from the WA State EBP Initiative

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Evidence-Based Practice Attitude Scale (EBPAS) | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Evidence-Based Practice Attitude Scale is a 15-item measure that captures a providers attitudes toward evidence-based practices. It consist subscales 1) appeal of EBP, 2) openness to new EBP, 3) likelihood of adopting an evidence-based practice, and 4) perceived divergence between current and evidence-based practices. The scores for the subscales range from 0 (not at all) to 4 (very great extent). The higher score equates to better attitude toward EBP.
Subjective Norms | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Subjective Norms Scale is based on Theory of Planned Bheavior (TBP) which consist of two implementation-related subject norms sub scales: descriptive norms and injuctive norms. Each subscale include four items with score ranging from -3 to 3, with positive scores reflective more descriptive and injunctive norms.
Outcome Expectancies | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Outcome expectanies is a one-item measure that assess provider's view of the outcome of implementing evidence-based practice to be positive or negative. The score ranges from 0, strongly disagree to 4, strongly agree. The higher the score, the positive the provider's outcome expectancy.
Action Self-Efficacy | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Action Self-Efficacy Scale is a modified version of the Teacher's Self-Efficacy Scale used to assess provider's confidence and self-efficacy in using the given evidence-based practice. This is 4-item measure with score ranging from 1, very false to 7, very true. The higher the score the more confidence the provider has in their ability to start using the evidence-based practice.
Maintenance Self-Efficacy | immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Maintenance Self-Efficacy measure is used to asses provider's confidence and self-efficacy in continuing to use the given evidence-based practice. It is a one item measure with score ranging from 1, very false to 7, very true. The higher the score the more confidence the provider has in their ability to continue using the evidence-based practice.
Perceived Needs | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Perceived Needs is a 1-item measure that assess if they have to improvie their skills in supporting students' mental health. The scores are 0- no, 1-I don't know, and 3-Yes.
Modified Intention to Implement Scale (MIIS) | Baseline, immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Modified Intentions to Implement Scale is used to understand a provider's intention to implement the given evidence-based practice. The survey includes 5-items, and the score ranges from -3, strongly disagree to 3, strongly agree.
Intervention Usability Scale (IUS) | immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Intervention Usability Scale (IUS) is a an 10-tem scale that assess the usability of evidence-based practice. The score ranges from 0, strongly disagree to 4, strongly agree. The higher score indicates that the provider finds the evidence-based practice is easier to use.
Action Plan | immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Action Plan is a one item measure to assess if the provider has an action plan in place to implement evidence-based practice. The score ranges from from 0, none are in place to 3, all are in place. The higher score, the more the provider has planned out evidence practice implementation.
Coping Plan | immediately after training, 2 weeks after training, 1 month after training, 2 months after training, 3 months after training
  Coping Plan is a one item measure to assess if the provider has come up with solutions to overcome any problems they face while implementing evidence-based practice. The score ranges from from 0, none are in place to 3, all are in place. The higher score, the more the provider has planned out evidence practice impementation.

SECONDARY OUTCOMES:
School Implementation Leadership Scale (S-ILS) | 2 weeks after training
  The School Implementation Leadership Scale (SILS) is an 25-item scale that assesses the degree to which a school's leader is perceived to engage in eight specific behaviors that are supportive of EBP implementation which both principals and educators complete. The eight subscales include: 1) supportive; 2) perseverant; 3) communication; 4) proactive; 5) availability; 6) knowledgeable; 7) vision/mission; and 8) distributed leadership.
School Implementation Climate Scale (S-ICS) | 2 weeks after training
  The School Implementation Climate Scale (SICS) is an 21-item scale for principals' and educators' shared perceptions of the policies, practices, and procedures that are expected, rewarded, and supported. The six subscales include: 1) focus on EBPs; 2) educational support for EBPs; 3) recognition for EBPs; 4) use of data to support EBPs; 5) existing supports to deliver EBPs; and 6) integration of EBPs.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No